CLINICAL TRIAL: NCT05324826
Title: Comparison of the Effectiveness of Handheld Ultrasound with MRI for Diagnosing Patients with Temporomandibular Joint Disorders
Brief Title: Effectiveness of Handheld Ultrasound for Diagnosing Patients with TMD
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Butterfly Network (Industry)
Responsible Party: Sponsor
Other Study IDs: B2022:010
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Joint Disorders; Magnetic Resonance Image; Handheld Ultrasound
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Butterfly Network handheld ultrasound — Patients would be examined with a handheld US machine which would allow for dynamic imaging chairside and could easily be integrated into both hospital-based and private clinical practices. This would allow the patient to benefit from realtime imaging and a faster preliminary diagnosis with virtually no additional risks.

SUMMARY:
The aim of this research is to add to the limited body of knowledge comparing the effectiveness of ultrasound (US) to MRI diagnoses in patients with TMJ disorders. More specifically, we will review the efficacy of handheld US devices, which has not yet been done to the author's knowledge.

DETAILED DESCRIPTION:
Currently, patients complaining of temporomandibular joint (TMJ) pain are evaluated clinically, which includes measurements of their maximal incisal opening (MIO) lateral and protrusive excursions, recording their current pain duration and frequency, and any clicking/popping/grinding of the joints. Based on these findings, the patient is sent for an MRI if temporomandibular joint disorder is suspected.

MRI is currently the gold standard of care for imaging of the joint, as it provides valuable information on the position, morphology and signal intensity of the joints and its surrounding structures. Magnetic resonance imaging (MRI) is currently the gold standard of imaging for diagnosis of internal derangement due to its ability to provide valuable information on the position, morphology and signal intensity of the joints and its surrounding structures. However, using MRI is not without its challenges, as patients with severe TMJ pain find it difficult to complete a full TMJ series and access to MRI is often restricted due to limited locations and associated waits, further prolonging time between initial consultation and diagnosis. In addition, MRI is contraindicated in patients with metallic implants, coronary and peripheral artery stents, cardiac pacemakers, prosthetic heart valves, intrauterine contraceptive devices, and claustrophobia. For these reasons, the author believes that attempting to find an alternative reliable screening tool for internal derangement is a worthwhile endeavor. For this study, handheld ultrasound would be used at the time of clinical examination to come up with a preliminary diagnosis, and this diagnosis would be compared to the MRI findings.

ELIGIBILITY:
Inclusion Criteria:

* The patient population will be those patients who meet the criteria for temporomandibular joint disorders based on clinical examination and patient history, including anterior disc displacement with or without reduction, joint effusion, or degenerative joint disease.

Exclusion Criteria:

* Patients under the age of 18.
* Patients unable to consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will be those patients who meet the criteria for temporomandibular joint disorders based on clinical examination and patient history, including anterior disc displacement with or without reduction, joint effusion, or degenerative joint disease. There is no requirement for a control group, because the preliminary diagnosis obtained from the ultrasound will be compared to the MRI results on the same patient.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the diagnosis obtained from handheld ultrasound to the diagnosis obtained from MRI | April 2022-December 2024
  Diagnosis obtained from handheld ultrasound will be compared to diagnosis obtained from MRI. This would include: anterior disc displacement with reduction, anterior disc displacement without reduction, joint effusion and osteoarthritic changes

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Shah, BDS, FRCDC, Study Director — University of Manitoba
Locations (1):
- Dr. Adnan Shah, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Friedman SN, Grushka M, Beituni HK, Rehman M, Bressler HB, Friedman L. Advanced Ultrasound Screening for Temporomandibular Joint (TMJ) Internal Derangement. Radiol Res Pract. 2020 May 4;2020:1809690. doi: 10.1155/2020/1809690. eCollection 2020. PMID 32426167
- [Background] Taskaya-Yilmaz N, Ogutcen-Toller M. Magnetic resonance imaging evaluation of temporomandibular joint disc deformities in relation to type of disc displacement. J Oral Maxillofac Surg. 2001 Aug;59(8):860-5; discussion 865-6. doi: 10.1053/joms.2001.25015. PMID 11474436
- [Background] Talmaceanu D, Lenghel LM, Bolog N, Popa Stanila R, Buduru S, Leucuta DC, Rotar H, Baciut M, Baciut G. High-resolution ultrasonography in assessing temporomandibular joint disc position. Med Ultrason. 2018 Feb 4;1(1):64-70. doi: 10.11152/mu-1025. PMID 29400370
- [Background] Kumar R, Pallagatti S, Sheikh S, Mittal A, Gupta D, Gupta S. Correlation Between Clinical Findings of Temporomandibular Disorders and MRI Characteristics of Disc Displacement. Open Dent J. 2015 Jul 31;9:273-81. doi: 10.2174/1874210601509010273. eCollection 2015. PMID 26464595
- [Background] Yilmaz D, Kamburoglu K. Comparison of the effectiveness of high resolution ultrasound with MRI in patients with temporomandibular joint disorders. Dentomaxillofac Radiol. 2019 Jul;48(5):20180349. doi: 10.1259/dmfr.20180349. Epub 2019 Feb 28. PMID 30810356